CLINICAL TRIAL: NCT03244605
Title: Clinical Study on the Effect of Comprehensive Rehabilitation Program on Quality of Life and Long-term Survival in Postoperative Non Small Cell Lung Cancer Patients
Brief Title: Efficacy Study of Comprehensive Rehabilitation Program in Postoperative NSCLC Patients
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Shanghai University of Traditional Chinese Medicine (Other)
Collaborators: Shanghai Chest Hospital (Other); Shanghai Pulmonary Hospital, Shanghai, China (Other); Shanghai Cancer Hospital, China (Other); Huadong Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SHUTCM001
Record Dates: First submitted 2017-07-19; First posted 2017-08-09 (Actual); Last update posted 2019-06-12 (Actual); Status verified 2019-04

CONDITIONS: Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Rehabilitation training plus TCM (Experimental): Rehabilitation training include aerobic exercise training and Liu Zi Jue lung exercises, which will be started in one month after operation.
  Prescriptions formulated into granules origin from Professor Xu Ling in Yueyang hospital. Package of granules is made into three types with functions such as benefiting Qi recipe, benefiting Yin recipe and detoxication and resolving masses recipe. Each package contained 20g of water-soluble herbal granules that were manufactured at a Good Manufacture Practice standard facility (Tian Jiang Ltd, Jiangyin, China). Each package was labeled with a serial number. The prescription form comprised the stock list with both the name and serial number.The patient will take TCM granules for 3 months.
  Interventions: Other: Rehabilitation Training; Drug: TCM
- Rehabilitation education plus placebo (Placebo Comparator): Patients who received rehabilitation education will not accept rehabilitation training.
  We compromise the raw materials for the placebo including food color and artificial flavors. The placebo and therapeutic packages were stored in different cabinets, and only the dispensing technician knew the contents of the packages.
  The patient will take placebo granules for 3 months.
  Interventions: Other: Rehabilitation Education; Drug: placebo

INTERVENTIONS:
Other: Rehabilitation Training — Patients will be trained in one month after operation. Rehabilitation training include aerobic exercise training (using cycle ergometer for 7-14 times at all, once a day, 15-20 min/time and using treadmill for 7-14 times at all, once a day, 15-20 min/time according to the patient's endurance) and Liu Zi Jue lung exercises, which strengthen the lung function of the human body in Chinese traditional health culture, five times a week, 15 min/time.
  Other Names: aerobic exercise training; Liu Zi Jue lung exercises
  Arms: Rehabilitation training plus TCM
Other: Rehabilitation Education — General health education
  Other Names: health education
  Arms: Rehabilitation education plus placebo
Drug: TCM — three types with functions such as benefiting Qi recipe, benefiting Yin recipe and detoxication and resolving masses recipe.
  Other Names: Prescriptions from Professor Xu Ling
  Arms: Rehabilitation training plus TCM
Drug: placebo — three types with functions such as benefiting Qi recipe, benefiting Yin recipe and detoxication and resolving masses recipe，with the same color, smell，taste weight and package
  Other Names: control
  Arms: Rehabilitation education plus placebo

SUMMARY:
The investigators performed a multi-centered, randomized, placebo-controlled, prospective clinical trial on the effect of comprehensive rehabilitation program to improve quality of life(QOL) and long-term survival of postoperative patients with early lung cancer. The investigators plan to enroll 236 cases in 3 years (118 cases for rehabilitation training plus traditional Chinese medicine (TCM), 118 cases for rehabilitation education plus placebo), expecting that comprehensive rehabilitation program has a better efficacy on improving QOL and long-term survival.

DETAILED DESCRIPTION:
Non-Small-Cell Lung Cancer（NSCLC）is one of the malignancies with high incidence and mortality. In recent years, surgery become the preferred treatment for early stage of NSCLC. Patients with stage IA-IIIA lung cancer can undergo radical surgery, but postoperative lung cancer patients also have shortness of breath, chest pain, cough, expectoration, upper limb dysfunction and other symptoms. The symptoms seriously affect the quality of life and follow-up treatment. Comprehensive rehabilitation program may alleviate the symptoms as an effective treatment which including rehabilitation training and TCM.

The investigators performed a multi-centered, randomized, placebo-controlled, prospective clinical trial on the effect of comprehensive rehabilitation program to improve quality of life(QOL) and long-term survival of postoperative patients who are not recommended for postoperative chemotherapy at stage IA and IB. Patients are randomized into observational group (rehabilitation training plus TCM), and control group (rehabilitation education plus placebo). The treatment should be last three months and the patients will be followed up regularly. The primary efficacy assessments are: (1) QOL (QLQ-LC43 scale); (2) Pulmonary function test(PFTs): 1) Forced vital capacity (FVC); 2) Forced expiratory volume in one second (FEV1); 3) Forced expiratory flow rate from 25% to 50% (FEF25-50); 4) Residual volume (RV); 5) Total lung capacity (TLC). Secondary efficacy assessments are: (1) 2 years disease-free survival; (2) TCM symptoms changes; (3) Tumer markers (CEA, CA-125 and CYFRA21-1); (4) Exercise tolerance; (5) Toxicity, side effects and security of the treatments will be assessed at the same time. The investigators plan to enroll 236 cases in 3 years (118 cases for rehabilitation training plus TCM, 118 cases for rehabilitation education plus placebo), expecting that comprehensive rehabilitation program has a better efficacy on improving QOL and long-term survival.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically or cytologically confirmed stage Ia-IIIa non small cell lung cancer;
* Between the ages of 18 to 75 years old;
* The score of ECOG ≥2 points
* Without major organ dysfunction: hemoglobin ≥10 g/dL, absolute neutrophil count (ANC) ≥1.5*10^9/L, platelets ≥100 *10^9/L; normal hepatic and renal function

Exclusion Criteria:

* Indefinite pathological diagnosis;
* Expected survival time < 6 months
* Combined with heart, liver, kidney and hematopoietic system and other serious diseases
* The patient was treated with antibiotics or infected one week before the test;
* Pregnant or child breast feeding women;
* Mental or cognitive disorders;

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 236 (Estimated)
Dates: Start 2016-10-01 (Actual); Primary Completion 2019-09-30 (Estimated); Study Completion 2019-12-30 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in Quality of life (QOL) | baseline, at 3 months
  QOL is assessed using European Organization for Research and Treatment of Cancer Quality of Life Questionnaire-Lung Cancer 43 (EORTC QLQ-LC43).

SECONDARY OUTCOMES:
Residual capacity (RV) | after intervention at 2 weeks
  RV is measured in a test known as Lung valume(LV)spirometry,a type of pulmonary function test.RV is the volume of air remaining in the lungs after a maximal expiratory effort.
Total lung capacity（TLC） | after intervention at 2 weeks
  TLC is measured in a test known as Lung valume(LV)spirometry,a type of pulmonary function test.TLC equals the vital capacity plus the residual capacity.
Forced vital capacity (FVC) | after intervention at 2 weeks
  FVC is the volume of air exhaled with maximum effort and speed after a full inspiration. FVC is measured in a test known as spirometry, a type of pulmonary function test.
Forced expiratory volume in one second(FEV1) | after intervention at 2 weeks
  FEV1 is an individual test measure used to assess limitations in airflow, a type of pulmonary function test,which measures the amount of air exhaled in onesecond.
Maximum mid expiratory flow(MMEF) | after intervention at 2 weeks
  MMEF is forced expiratory flow between 25% and 75% of forced vital capacity,a type of pulmonary function test.
Disease-free survival (DFS) | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 60 months
  Time from randomization to first recurrence or metastasis
TCM symptoms changes | after intervention at 3 months
  TCM symptoms changes are according to the lung cancer symptom classification quantization table in "Guiding Principles for Clinical Research of Traditional Chinese Medicine in the Treatment of Lung Cancer (2002 Edition)"
Tumor markers | after intervention at 3 months
  Tumor markers include CEA, CA-125 and CYFRA21-1
Safety assessment evaluated according to Common Toxicity Criteria | after intervention at 3 months
  Safety assessment is evaluated according to Common Toxicity Criteria (CTC 3.0)

CONTACTS AND LOCATIONS:
Overall Officials: Ling Xu, MD & PhD, Principal Investigator — Shanghai University of Traditional Chinese Medicine
Locations (1):
- YueYang Hosptial of Intergrated Traditional Chinese and Western Medicine,Shanghai University of Traditional Chinese Medicine, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Qin X, Bi L, Yang W, He Y, Gu Y, Yang Y, Gong Y, Wang Y, Yan X, Xu L, Xiao H, Jiao L. Dysbiosis of the Gut Microbiome Is Associated With Histopathology of Lung Cancer. Front Microbiol. 2022 Jun 14;13:918823. doi: 10.3389/fmicb.2022.918823. eCollection 2022. PMID 35774470